CLINICAL TRIAL: NCT06297941
Title: A Phase 1, Multicenter, Open-Label Study of REM-422, an MYB mRNA Degrader, in Patients With Relapsed/Refractory AML or Higher-Risk MDS
Brief Title: Study of REM-422 in Patients With AML or Higher Risk MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Remix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REM-422-102
Record Dates: First submitted 2024-02-23; First posted 2024-03-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes; Higher Risk Myelodysplastic Syndromes; Acute Myeloid Leukemia; Acute Myeloid Leukemia Refractory
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REM-422 (Experimental): Dose Escalation: Participants will receive escalating doses of REM-422 to determine Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D)-422, oral capsule administered once daily
  Dose Expansion: Participants will receive REM-422 at the identified RP2D Treatment will continue until disease progression, therapy intolerance, or participant withdrawal Safety evaluation will continue until 30 days of last administration of REM-422
  Interventions: Drug: REM-422

INTERVENTIONS:
Drug: REM-422 — REM-422 is a first in class, small molecule mRNA inhibitor that reduces expression of the MYB transcription factor
  REM-422 will be administered orally once daily

SUMMARY:
The goal of this study is to determine the safety and antitumor effects of REM-422, a MYB mRNA degrader, in people with Higher Risk MDS and relapsed/refractory AML

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, multicenter study investigating REM-422, a potent, selective, and oral small molecule mRNA degrader that reduces expression of the MYB transcription factor for patients with higher risk MDS or relapsed/refractory AML.

This study includes a Dose Escalation Phase and a Dose Expansion Phase. The purpose of the Dose Escalation Phase is to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of REM-422 in patients with higher risk MDS or relapsed/refractory AML. The purpose of Dose Expansion is to further evaluate the safety and anti-tumor activity of the RP2D carried forward from Dose Escalation.

Participation in this study will continue until disease progression, therapy intolerance, or participant withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide informed consent.
2. Be 18 or older at the time of informed consent.
3. Disease criteria:

   Histologically confirmed diagnosis of either:
   1. R/R AML, defined as relapse after transplantation, second or later relapse, refractory to initial induction or reinduction treatment or to initial treatment with hypomethylating (HMA)-based combinations, relapse after initial treatment, or otherwise considered relapsed or refractory in the opinion of the Investigator.
   2. High-risk and very-high-risk (VHR) MDS (higher-risk) per the International Prognostic Scoring System-Revised (IPSS-R) and/or International Prognostic Scoring System-Molecular (IPSS-M).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Has agreed to undergo serial blood and bone marrow sampling.
6. Participants must have completed systemic non-investigational therapy at least 14 days prior to initiating REM-422. Hydroxyurea is permissible for controlling peripheral leukemic blasts prior to enrollment and for up to 28 days following initiation of REM-422.
7. Toxicities from prior therapy must be either stable or recovered to ≤ Grade 1.
8. Participants must be able to swallow and retain oral medications.
9. Oxygen saturation > 92% on room air or up to 2 L/min supplemental oxygen by nasal cannula with ≤ Grade 1 dyspnea.
10. People of childbearing potential (POCBP) must have a negative serum beta-human chorionic gonadotropin test result.
11. POCBP must agree to use acceptable, effective methods of contraception and not donate ova from screening until 6 months after discontinuation of REM-422. Women who have undergone surgical or ablative sterilization or who have been postmenopausal for ≥ 2 years are not considered to be of childbearing potential.
12. Men must agree to use acceptable, effective methods of contraception and must agree not to donate sperm from the start of receiving REM-422 until 6 months after discontinuation of REM-422.
13. Adequate organ function and laboratory parameters

Exclusion Criteria:

1. Active central nervous system (CNS) leukemia or a confirmed diagnosis of CNS leukemia.
2. Has undergone hematopoietic stem cell transplantation (HSCT) within 60 days of the first dose of REM-422 or is receiving immunosuppressive therapy post HSCT at the time of screening, or has GVHD requiring systemic treatment (topical steroids for ongoing skin GVHD is permitted).
3. Has immediate, life-threatening, severe complications of leukemia, such as uncontrolled bleeding, pneumonia with hypoxia or sepsis, and/or disseminated intravascular coagulation.
4. Known hypersensitivity or contraindication to any component of REM-422 or to drugs chemically related to REM-422 or its excipients.
5. Clinically significant active infection. Note: Patients with simple urinary tract infection or uncomplicated bacterial pharyngitis responding to active treatment are permitted. Note: Patients receiving intravenous (IV) antibiotics ≤ 7 days prior to enrollment are excluded (prophylactic antibiotics, antivirals, or antifungals are permitted).
6. Evidence of active HIV infection.
7. Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
8. Primary immunodeficiency.
9. Current or expected need for daily systemic corticosteroid therapy ≥ 10 mg of prednisone equivalent.

   Note: Patients who are receiving topical or inhaled corticosteroids with minimal systemic absorption are eligible for enrollment and may continue with minimal corticosteroid use as long as they are on a stable dose.
10. Live vaccine ≤ 6 weeks prior to the start of REM-422.
11. Use of strong CYP3A inhibitors (except azole antifungals) or CYP3A inducers
12. Drugs that reduce gastric acidity, such as H2-receptor antagonists (eg, ranitidine, famotidine) and proton pump inhibitors (eg, omeprazole, esomeprazole) within 7 days prior to the initiation of REM-422 administration or during the study.
13. Currently pregnant, have intentions to become pregnant during the study duration, or are currently lactating.
14. Has dysphagia, short-gut syndrome, gastroparesis, or any other condition that limits the ingestion or gastrointestinal absorption of orally administered drugs.
15. Current use of prohibited medication ≤ 1 week before starting REM-422.
16. Clinically significant cardiovascular disease:
17. Has undergone major surgery (opening a mesenchymal barrier such as the pleural cavity, peritoneum, or meninges or surgical procedures requiring general anesthesia) < 4 weeks prior to enrollment.
18. History of organ transplant that requires use of immunosuppressive agents.
19. History or current autoimmune disease requiring systemic treatment (eg, Crohn's disease, ulcerative colitis, rheumatoid arthritis, systemic lupus).
20. Radiation therapy ≤ 7 days prior to the start of REM-422.
21. Concurrent or previous other malignancy ≤ 2 years of enrollment, except curatively treated malignancies including basal or squamous cell skin cancer, breast cancer, prostate intraepithelial neoplasm, and carcinoma in situ of the cervix.
22. Receiving any other investigational treatment for any indication ≤ 3 weeks prior to enrollment.
23. Unwillingness or inability to follow protocol requirements.
24. Any condition that, in the opinion of the Investigator, would interfere with evaluation of REM-422 or interpretation of the participant's safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Treatment Emergent Adverse Events (TEAEs) | 24 months
  Frequency and severity of Treatment Emergent Adverse Events (TEAEs) will be evaluated according to the NCI-CTCAE version 5.0 and number of participants with Dose Limiting Toxicities will be assessed to determine Safety and Tolerability of REM-422 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | Assessed at the end of Cycle 1 (each cycle is 28 days) for each participant for approximately 24 months
  Frequency and severity of Treatment Emergent Adverse Events (TEAEs) will be evaluated according to the NCI-CTCAE version 5.0 and the number of participants with Dose Limiting Toxicities will be assessed from the date of first dose of REM-422 until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months

SECONDARY OUTCOMES:
AML: Rate of Complete Response (remission) (CR) | 24 months
  Rate of Complete Response (CR) will be measured based on Investigator assessment per the modified International Working Group (IWG) response criteria 2003 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
AML: Rate of CR with partial hematologic recovery (CRh) | 24 months
  Rate of Complete Response (CR) with partial hematologic recovery (CRh) will be measured based on Investigator assessment per the modified International Working Group (IWG) response criteria 2003 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
AML: Duration of CR | 24 months
  Duration of CR will be evaluated per the modified International Working Group (IWG) response criteria 2003 following treatment with REM-422 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
AML: Duration of CRh | 24 months
  Duration of CRh will be evaluated per the modified International Working Group (IWG) response criteria 2003 following treatment with REM-422 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
AML: Overall response rate (ORR) (CR + CRh + CRi + PR) with incomplete hematologic recovery [CRi] + partial response [PR]) per modified IWG response criteria 2003 based on Investigator assessment | 24 months
  Duration of Overall Response Rate (ORR) will be evaluated per the modified International Working Group (IWG) response criteria 2003 following treatment with REM-422 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
AML: Duration of response (DOR) | 24 months
  Duration of Response (DoR) will be evaluated following treatment with REM-422 based on Investigator assessment for participants who achieve a response per IWG response criteria 2003, defined as the time from when response criteria are first met for CR, CRi, CRh, or PR until progressive disease (PD) per IWG response criteria 2003 is documented or death, whichever occurs first
MDS: Rate of Compete Response (CR) | 24 months
  Rate of CR will be evaluated based on Investigator assessment per IWG 2023 response criteria following treatment with REM-422 for participants who achieve a Complete Response (CR), defined as the time from when criteria are first met for CR until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
MDS: Duration of Complete Response (CR) | 24 months
  Duration of CR will be evaluated per IWG 2023 response criteria following treatment with REM-422 based on Investigator assessment for participants who achieve a CR per IWG response criteria 2003, defined as the time from when response criteria are first met for CR until progressive disease (PD) per IWG response criteria 2003 is documented or death, whichever occurs first
MDS: Overall Response Rate (ORR) | 24 months
  ORR will be evaluated per IWG 2023 response criteria based on Investigator assessment following treatment with REM-422 from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 24 months.
MDS: Duration of Response (DOR) | 24 months
  DOR will be evaluated following treatment with REM-422 based on Investigator assessment for participants who achieve a response per IWG 2023 response criteria, defined as the time from when criteria are first met for CR, CRi, CRh, or PR until PD per IWG 2023 or death, whichever occurs first
Determine pharmacokinetic profile (Cmax) of REM-422 | 24 months
  Measure Maximal concentration (Cmax) of REM-422
Determine pharmacokinetic profile (Cmin) of REM-422 | 24 months
  Measure Minimal concentration (Cmin) of REM-422
Determine pharmacokinetic profile (Tmax) of REM-422 | 24 months
  Measure Time to peak drug concentration (Tmax) of REM-422
Determine pharmacokinetic profile (AUC) of REM-422 | 24 months
  Measure Area Under the Curve (AUC) of REM-422

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowden, MD, Study Chair — Remix Therapeutics
Locations (9):
- United States (5):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- France (4):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - AP-HP - Hôpital Saint-Louis, Paris
  - IUCT-Oncopole, Toulouse
  - Institut de Cancerologie Gustave-Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No